CLINICAL TRIAL: NCT01657032
Title: Efficacy of Lactobacillus GG With Diosmectite in Treatment Children With Acute Gastroenteritis: A Double Blind Randomized, Placebo- Controlled Trial
Brief Title: Efficacy of Lactobacillus GG With Diosmectite in Treatment Children With Acute Gastroenteritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KB2010
Record Dates: First submitted 2012-07-05; First posted 2012-08-03 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2010-01

CONDITIONS: Diarrhea
Keywords: diarrhea; probiotics; diosmectite
MeSH Terms: conditions — Diarrhea | interventions — Smectite; smecta; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus GG and Smectite (Experimental): Children received:
  * LGG (ATCC 53103), dose 6×10 9 colony forming units (CFU), once a day for 7 days and
  * smectite, dose 3 g, once daily orally until diarrhea stopped
  Interventions: Dietary Supplement: Smectite; Dietary Supplement: Lactobacillus GG
- Lactobacillus GG and Placebo (Placebo Comparator): Children received:
  * LGG (ATCC 53103), dose 6×10 9 colony forming units (CFU), once a day for 7 days and
  * placebo (glucose), dose 3 g, once daily orally until diarrhea stopped
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Lactobacillus GG

INTERVENTIONS:
Dietary Supplement: Smectite — Eligible children received smectite (3g) once a day till diarrhea stop with LGG (ATCC 53103) at a daily dosage of 6×10 9 colony forming units (CFU) in one dose for 7 days.
  Other Names: Smecta
  Arms: Lactobacillus GG and Smectite
Dietary Supplement: Placebo — Eligible children received placebo: glucose (3g) once a day till diarrhea stop with LGG (ATCC 53103) at a daily dosage of 6×10 9 colony forming units (CFU) in one dose for 7 days.
  Other Names: glucose
  Arms: Lactobacillus GG and Placebo
Dietary Supplement: Lactobacillus GG — All children received LGG (ATCC 53103), dose 6×10 9 colony forming units (CFU), once a day for 7 days with placebo or smectite
  Other Names: Dicoflor 30

SUMMARY:
Treatment diarrhea with Lactobacillus GG or smectite has proven efficacy. A randomized, double blind, placebo-control trial was performed to assess the effectiveness of both LGG and smectite in management of children with acute gastroenteritis (AGE).

DETAILED DESCRIPTION:
ESPGHAN agreed to use probiotics, with proven efficacy, and smectite in treatment of AGE as an adjunct to standard rehydration therapy. Among probiotics Lactobacillus GG were found to be beneficial in meta-analyses. Treatment with LGG was associated with a significant reduction in diarrhea duration.

A recent review systematically evaluated the efficacy of smectite in treating acute infections diarrhea in infants and children.

ELIGIBILITY:
Inclusion Criteria:

* children < 5 years old
* diarrhea (defined as the passage of 3 or more loose or watery stools per day) for > 1 day but < 5 days
* inform consent sing

Exclusion Criteria:

* diarrhea < 1 or > 5 days,
* a recent history of diarrhea indicated either by parents/guardian or hospital case notes,
* underlying chronic gastrointestinal disease,
* undernutrition (weight/height ratio below the 5th percentile),
* systematic infection,
* immune defects or immunosuppressive treatment

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatrics, The Medical University of Warsaw, Warsaw, Warsaw, Poland

REFERENCES:
- [Background] Guarino A, Albano F, Ashkenazi S, Gendrel D, Hoekstra JH, Shamir R, Szajewska H; ESPGHAN/ESPID Evidence-Based Guidelines for the Management of Acute Gastroenteritis in Children in Europe Expert Working Group. European Society for Paediatric Gastroenterology, Hepatology, and Nutrition/European Society for Paediatric Infectious Diseases evidence-based guidelines for the management of acute gastroenteritis in children in Europe: executive summary. J Pediatr Gastroenterol Nutr. 2008 May;46(5):619-21. doi: 10.1097/MPG.0b013e31816e219e. No abstract available. PMID 18493225
- [Background] Guarner F, Schaafsma GJ. Probiotics. Int J Food Microbiol. 1998 Feb 17;39(3):237-8. doi: 10.1016/s0168-1605(97)00136-0. No abstract available. PMID 9553803
- [Background] Szajewska H, Skorka A, Ruszczynski M, Gieruszczak-Bialek D. Meta-analysis: Lactobacillus GG for treating acute diarrhoea in children. Aliment Pharmacol Ther. 2007 Apr 15;25(8):871-81. doi: 10.1111/j.1365-2036.2007.03282.x. PMID 17402990
- [Background] Szajewska H, Dziechciarz P, Mrukowicz J. Meta-analysis: Smectite in the treatment of acute infectious diarrhoea in children. Aliment Pharmacol Ther. 2006 Jan 15;23(2):217-27. doi: 10.1111/j.1365-2036.2006.02760.x. PMID 16393300

RESULTS

PARTICIPANT FLOW:
Groups:
- Lactobacillus GG and Smectite: Children received:
  * LGG (ATCC 53103), dose 6×10 9 colony forming units (CFU), once a day for 7 days and
  * smectite, dose 3 g, once daily orally until diarrhea stopped
  Smectite: Eligible children received smectite (3g) once a day till diarrhea stop with LGG (ATCC 53103) at a daily dosage of 6×10 9 colony forming units (CFU) in one dose for 7 days.
  Lactobacillus GG: All children received LGG (ATCC 53103), dose 6×10 9 colony forming units (CFU), once a day for 7 days with placebo or smectite
- Lactobacillus GG and Placebo: Children received:
  * LGG (ATCC 53103), dose 6×10 9 colony forming units (CFU), once a day for 7 days and
  * placebo (glucose), dose 3 g, once daily orally until diarrhea stopped
  Placebo: Eligible children received placebo: glucose (3g) once a day till diarrhea stop with LGG (ATCC 53103) at a daily dosage of 6×10 9 colony forming units (CFU) in one dose for 7 days.
  Lactobacillus GG: All children received LGG (ATCC 53103), dose 6×10 9 colony forming units (CFU), once a day for 7 days with placebo or smectite
Period: Overall Study
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo
Started | 44 | 44
Completed | 44 | 37
Not Completed | 0 | 7
Not completed — Lost to Follow-up | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 17.5 [10.0 to 22.5] | 18 [11 to 30] | 18 [10 to 23]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44 | 44 | 88
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 15 | 38
  Male | 21 | 29 | 50
Region of Enrollment [Number; unit: participants]
  Poland | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: Duration of Diarrhea
Description: The primary outcome measure is duration of diarrhea (counted in days; from the first loose stool to the last one; end of diarrhea defined as last loose stool or at least 12hours without stool).
Time Frame: counted in days during 7days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo
Number analyzed (Participants) | 44 | 37
days | 2 [1 to 3] | 2 [1 to 2]
Statistical Analysis 1: Comparison: Lactobacillus GG and Smectite; Test type: Non-Inferiority or Equivalence — The differences between the study groups were considered significant when the P value was <0.05; p = 0.43, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Frequency of Loose Stools,
Description: number of loose stools during 7 days
Time Frame: number of loose stools during 7 days
Measure: Median (Inter-Quartile Range); unit: number of loose stools during 7days
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo
Number analyzed (Participants) | 44 | 37
number of loose stools during 7days | 10.5 [5 to 21] | 10 [5 to 15]

3. Secondary Outcome: Consistency of Stools
Description: consistency of stools using Bristool Stool Scale Form on day 4-th. (The Bristol stool scale form is a medical aid designed to classify the form of human faeces into seven categories.
  Type 1 Separate hard lumps, like nuts (hard to pass) Type 2 Sausage-shaped but lumpy Type 3 Like a sausage but with cracks on the surface Type 4 Like a sausage or snake, smooth and soft Type 5 Soft blobs with clear-cut edges Type 6 Fluffy pieces with ragged edges, a mushy stool Type 7 Watery, no solid pieces. Entirely liquid Types 1-2 indicate constipation, with 3 and 4 being the ideal stools (especially the latter), as they are easy to defecate while not containing any excess liquid, and 5, 6 and 7 tending towards diarrhoea.
Time Frame: day 4-th
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo
Number analyzed (Participants) | 44 | 37
Units on a scale | 5 [3 to 6] | 4 [0 to 5]

4. Secondary Outcome: Need for Antibiotic Therapy,
Description: need for antibiotic therapy because of diarrhea
Time Frame: yes/no, for 7days
Measure: Number; unit: participants
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo
Number analyzed (Participants) | 44 | 37
participants | 0 | 0

5. Secondary Outcome: Vomiting
Description: If the child vomiting after randomization (yes/no)
Time Frame: yes/no, for 7days
Measure: Number; unit: participants
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo
Number analyzed (Participants) | 44 | 37
participants | 9 | 11

6. Secondary Outcome: Vomiting
Description: How many times the child was vomiting (during the study)
Time Frame: how many times for 7days
Measure: Median (Inter-Quartile Range); unit: vomiting episodes
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo
Number analyzed (Participants) | 44 | 37
vomiting episodes | 0 [0 to 1] | 0 [0 to 0]

7. Secondary Outcome: Diarrhea Recurrence
Description: If the was a diarrhea recurrence during 7days
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo
Number analyzed (Participants) | 44 | 37
participants | 3 | 3

8. Secondary Outcome: Tolerance of Products
Description: tolerance of products (whether the child took medicaments),
Time Frame: 7days
Measure: Number; unit: participants
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo
Number analyzed (Participants) | 44 | 37
participants | 34 | 32

9. Secondary Outcome: Need for Hospitalization
Description: If the child need to hospitalized
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo
Number analyzed (Participants) | 44 | 37
participants | 34 | 31

10. Secondary Outcome: Need for Intravenous Therapy
Description: need for intravenous rehydration therapy (yes/no)
Time Frame: yes/no, for 7days
Measure: Number; unit: participants
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo
Number analyzed (Participants) | 44 | 37
participants | 23 | 25

11. Secondary Outcome: Duration of Intravenous Therapy
Description: need for intravenous rehydration therapy (how long if needed)
Time Frame: 7days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo
Number analyzed (Participants) | 44 | 37
days | 1 [0 to 1] | 1 [0 to 3]

ADVERSE EVENTS:
Time Frame: 7days
Arm/Group | Lactobacillus GG and Smectite | Lactobacillus GG and Placebo
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/37
Other Adverse Events (participants affected / at risk) | 0/44 | 0/37

LIMITATIONS AND CAVEATS:
A potential limitation of our study is the lack of perfect blinding. Patients received smectite or placebo in identical packages from the hospital pharmacy. After being dissolved in water, they were of different colors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes